CLINICAL TRIAL: NCT00891553
Title: Study CR9112792, a Study to Assess Bone Mineral Density Changes in Post-menopausal Osteoporotic Women Following Discontinuation of Ronacaleret or Placebo Treatment in Study CR9108963
Brief Title: CR9112792, a Follow-up of Study CR9108963
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112792
Record Dates: First submitted 2009-04-23; First posted 2009-05-01 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Osteoporosis
Keywords: bone mineral density; calcium-sensing receptor antagonist; ronacaleret; postmenopausal osteoporosis
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ronacaleret: Subjects receiving ronacaleret (200mg,300mg or 400mg) in study CR9108963 will be enrolled into this study.
  Interventions: Procedure: DXA
- Placebo: Subjects receiving placebo in study CR9108963 will be enrolled into this study.
  Interventions: Procedure: DXA

INTERVENTIONS:
Procedure: DXA — CR9112792 is a follow-up study of CR9108963, in which the effects of ronacaleret (100mg, 200mg, 300mg, 400mg) on bone mineral density (BMD), safety and tolerability were evaluated in comparison with placebo and 2 active comparators, alendronate and teriparatide. In this study we will follow-up subjects between 6 and 12 months after they discontinued treatment with placebo or ronacaleret (200mg, 300mg, 400mg) to evaluate the potential for mineralization of bone following cessation of ronacaleret therapy, evaluating lumbar spine and hip BMD by DXA. There is no administration of drug in this study.

SUMMARY:
The purpose of this study is to determine whether bone mineral density has increased in a subgroup of postmenopausal osteoporotic women from study CR9108963, between 6 and 12 months following cessation of ronacaleret therapy.

DETAILED DESCRIPTION:
CR9112792 is a follow-up study of CR9108963, the 12 month dose ranging study of ronacaleret (SB-751689), a calcium sensing receptor antagonist, in postmenopausal women with osteoporosis. CR9108963 evaluated the effects of ronacaleret (100mg, 200mg, 300mg, 400mg) on bone mineral density (BMD), safety and tolerability in comparison with placebo and 2 active comparators, alendronate and teriparatide. CR9108963 was terminated earlier than planned due to an observed lack of efficacy in lumbar spine and hip BMD. In this study we will follow-up subjects between 6 and 12 months after they discontinued treatment with ronacaleret to evaluate the potential for mineralization of bone following cessation of ronacaleret therapy. Subjects at pre-specified sites from the CR9108963 placebo, 200mg, 300mg and 400mg dose groups will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: Subject is willing and able to provide written informed consent.
* Subjects: Subjects must have completed through the Month 12 visit of study CR9108963, or have had an early withdrawal visit on or after their Month 10 visit.
* DXA: Subjects must have either a final evaluable spine or hip DXA scan in CR9108963 as confirmed by Synarc, taken within 4 weeks of the last dose of study medication.
* Study medication: Subjects must have been on placebo or ronacaleret 200mg, 300mg or 400mg for ≥299 days in study CR9108963.

Exclusion Criteria:

* Any treatment with a PTH-based therapy or strontium ranelate after discontinuation of treatment in study CR9108963.
* Chronic systemic corticosteroid [e.g., glucocorticoid, mineralocorticoid] treatment of more than 2 intra-articular injections within the past year or use of oral, parenteral, or long-term, high-dose inhaled corticosteroids. Treatment with any topical corticosteroid will not exclude the subject from participating.
* Treatment with any topical corticosteroid will not exclude the subject from participation.
* Treatment with fluoride (dose greater than 10mg/day) for osteoporosis after discontinuation of treatment in study CR9108963.
* Administration of any investigational drug after discontinuation of treatment in study CR9108963.
* Subject who, in the opinion of the investigator, is unfit for this study or unable to comply with the requirements of the protocol.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population for CR9112792 will include approximately 145 postmenopausal women of those enrolled in study CR9108963, identified from subjects willing to participate and meeting eligibility criteria at pre-specified sites.
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Percent change in BMD, as measured by DXA, at the lumbar spine (L1-L4) | 6 to 12 months from the final CR9108963 DXA to the CR9112792 study visit

SECONDARY OUTCOMES:
Percent change in BMD, as measured by DXA, at the total hip, trochanter and femoral neck | 6 to 12 months from the final CR9108963 DXA to the CR9112792 study visit
Percent change in BMD, as measured by DXA, at the lumbar spine (L1-L4) and total hip, trochanter and femoral neck | 16 to 25 months from the screening CR9108963 DXA to the CR9112792 study visit
Percent change in BMD, as measured by DXA, at the lumbar spine (L1-L4) and total hip, trochanter and femoral neck | 12 to 18 months from the month 6 CR9108963 DXA to the CR9112792 study visit

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Ballerup Municipality, Denmark
- Norway (2):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Hamar